CLINICAL TRIAL: NCT01933750
Title: A Prospective, Multicenter, Controlled Clinical Study of the PresVIEW Scleral Implant for the Improvement of Near Visual Acuity in Presbyopic Patients
Brief Title: Trial of the PresView Implant for the Improvement of Near Vision in Presbyopic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Refocus Ocular Europe, B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU-001; NCT01910207 (obsolete NCT alias)
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Presbyopia
Keywords: Presbyopia; Reading Glasses; Near Vision
MeSH Terms: conditions — Presbyopia; Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Randomized/Control (No Intervention): 7 patients randomized to deferred treatment/control cohort at the 3 sub-study control sites = 21
- Non-Randomized/Treatment (Experimental): Patients are non-randomized and if meet inclusion criteria receive the implantation of the PresVIEW device
  Interventions: Device: PresVIEW Device Implantation

INTERVENTIONS:
Device: PresVIEW Device Implantation
  Arms: Non-Randomized/Treatment

SUMMARY:
Study to determine the effectiveness of the PresVIEW Scleral Implant to improve near vision in patients who require reading glasses

ELIGIBILITY:
Inclusion Criteria:

* Age 45 or older at commencement of study
* Best Corrected Distance Visual Acuity of .80 (20/25) or better
* Patients must be alert, mentally competent, and able to comply with clinical study requirements

Exclusion Criteria:

* Any previous eye surgeries including cataract, LASIK (laser in situ keratomileusis), or eye muscle surgery
* Any chronic systemic diseases such as diabetes, heart disease, Lupus, etc.
* Any eye diseases such as eye inflammation, infection, cataract, or retinal diseases

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Near Visual Acuity | 12 Months
  Measurement of the distance Corrected Near Visual Acuity at 40 centimeters compared to baseline measurement. A minimum of 75% of patients with a bilateral post-operative Distance Corrected Near Visual Acuity of .5 (20/40) or better at 12 months

SECONDARY OUTCOMES:
Uncorrected Near Visual Acuity | 12 Months
  The percent of patients with a bilateral post-operative uncorrected near visual acuity (UCNVA) at 40 centimeters of .5 (20/40) or better at 12 months
Presence of Significant Safety Events | 24 months
  Several indicators of safety are monitored including but not limited to Best Corrected Distance Visual Acuity, Intra-ocular Pressure, and Chronic Inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- Midland Eye, Birmingham, United Kingdom